CLINICAL TRIAL: NCT04507477
Title: Ex-vivo Delivery of Rituximab to Prevent Post-transplant Lymphoproliferative Disease in Epstein-Barr Virus Mismatch Lung Transplant Recipients: A Pilot Trial
Brief Title: Ex-vivo Delivery of Rituximab to Prevent PTLD in EBV Mismatch Lung Transplant Recipients: A Pilot Trial
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19-6260
Record Dates: First submitted 2020-08-04; First posted 2020-08-11 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2021-07

CONDITIONS: Epstein-Barr Virus Infections; Post-transplant Lymphoproliferative Disorder
Keywords: Rituximab; EBV; EVLP; lung transplant
MeSH Terms: conditions — Epstein-Barr Virus Infections | interventions — Rituximab

STUDY DESIGN:
Intervention Model Description: At our institution, approximately 50% of donor lungs are put on ex-vivo lung perfusion (EVLP) for clinical purposes. If a patient consents to participate in this study and their donor is EBV positive, the donor lungs will first be put on EVLP. Rituximab will be administered to the donor lungs while they are on EVLP for 3 to 4 hours before the transplant is done in order to reduce the amount of EBV virus. The amount of time the donor lungs are on EVLP will not be changed as a result of participating in this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rituximab + Ex-vivo lung perfusion (Experimental): Donor lungs deemed suitable for such patients will undergo ex vivo lung perfusion (EVLP) as per standard practice. In clinical practice almost all adult donor lungs are EBV seropositive. If in the rare case the donor lung is EBV seronegative, then the lung transplant candidate/recipient will no longer need to be part of the study. Therefore, for EBV seropositive lungs meant for an EBV seronegative recipient, one dose of rituximab (500mg) will be added to the EVLP perfusate and be allowed to circulate for 3-4 hours. Lungs will then be transplanted as per standard procedure.
  Interventions: Biological: Rituximab

INTERVENTIONS:
Biological: Rituximab — For EBV seropositive lungs meant for an EBV seronegative recipient, one dose of rituximab (500mg) will be added to the EVLP perfusate and be allowed to circulate for 3-4 hours.
  Other Names: Rituxan

SUMMARY:
Post-transplant lymphoproliferative disorders (PTLD) can present as a type of malignancy that limits patient and graft survival after solid organ transplantation. Many early PTLDs are driven by the Epstein-Barr Virus (EBV).

Once acquired, EBV virus establishes latency in B-cells and can reactivate under immunosuppression. The highest risk transplant type to develop PTLD are lung transplants who have newly acquired EBV from their donors (D+/R-). There are no good modalities to prevent PTLD from developing after transplant. Rituximab is a monoclonal antibody that depletes B-cells thereby also reducing the burden of EBV. However, rituximab can have toxicities when given intravenously including infusion reactions and increased risk of reactions.

Furthermore, more than one dose is usually required. The Toronto Transplant program has developed a technology called ex vivo lung perfusion that repairs lungs outside of the body. Preliminary work has shown that rituximab given through the EVLP circuit can coat B-cells. We have also shown that there is no toxicity to the lung by giving rituximab. The current highly novel study proposes to treat donor lungs ex-vivo with rituximab in order to decrease the amount of B-cells and EBV in the graft. These lungs will then be transplanted into EBV negative patients with the hope that transmission of EBV would be reduced or prevented. Ten patients will be included in the current trial. Outcomes include safety, EBV viral load, and B-cell measurements in biopsies.

DETAILED DESCRIPTION:
Previous studies have shown that EBV D+/R- lung transplant patients have a high rate of post-transplant lymphoproliferative disease up to 22%. Various methods have been proposed to decrease the risk of PTLD in EBV D+/R- organ transplants. These include a) antiviral prophylaxis with valganciclovir; b) EBV viral load monitoring and reduction of immunosuppression; c) avoidance of polyclonal antibody induction; d) treatment of EBV viremia with ganciclovir +/- intravenous immunoglobulin; e) pre-emptive systemic rituximab for EBV viremia. Antiviral strategies which include (val)ganciclovir in particular do not have proven efficacy in this setting. In addition, current antivirals do NOT target latent virus which would be the predominant form of virus in the allograft, and is also the predominant viral state that drives B-cell proliferation. Rituximab is a chimeric monoclonal antibody that targets CD20+ B-cells. It has been used clinically for many years to treat a variety of diseases and is used in transplantation for induction. Rituximab has been used successfully as a prophylactic and therapeutic drug for the reduction of EBV viremia and PTLD in hematopoietic stem cell transplant recipients. Ex-Vivo Lung Perfusion (EVLP) is a novel method of donor lung preservation and treatment developed in Toronto which allows donor lungs to be treated for up to 12h or more under protective physiological conditions. This essentially creates a critical time window in which donor lungs can be optimally repaired prior to transplant. An advantage of ex-vivo delivery of rituximab includes the ability to deliver high-doses locally to the graft while potentially avoiding serious adverse effects in the recipient. Pre-clinical studies have shown that adding rituximab to the perfusate allows for safe delivery of the drug directly to the lungs and adjacent lymph nodes and is non-toxic. EBV D+/R- lung transplant patients have a high rate of PTLD. There are no proven prevention measures. Rituximab is a commonly used medication in transplant patients as well as for other indications. Rituximab depletes B cells in lung tissues and may reduce the transmission of EBV, thereby preventing PTLD. Giving Rituximab directly to the lungs will avoid systemic toxicity in the patient. The investigators hypothesize that donor lungs treated with Rituximab during ex vivo lung perfusion will result in B-cell depletion and therefore be less likely to transmit EBV, thereby reducing the risk of PTLD in the lung recipient. As noted above the advantages of delivering rituximab ex vivo include prevention of adverse effects of rituximab including systemic depletion of B-cells, reduced systemic immunosuppression, and infusion-related toxicities, and ability to deliver a high-dose locally to the allograft.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* Listed for single or double lung transplantation
* EBV (EBNA IgG and/or VCA IgG) seronegative (tested within the last 12 months)

Exclusion Criteria:

* EBV seropositivity at any time prior to transplant
* History of Cancer (eg, lymphoma)
* History of receiving rituximab or allergy to rituximab
* Underlying immunodeficiency (eg, common variable immune deficiency)
* Unable or unwilling to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-07-07 (Actual); Primary Completion 2022-12-07 (Estimated); Study Completion 2023-02-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Primary Graft Dysfunction | 1 week post-transplant
  Primary graft dysfunction (PGD) will be measured using previously defined criteria: PGD2 will be a PaO2:FiO2 of 200-300 mmHg with pulmonary edema on chest radiograph whereas PGD3 will be a PaO2:FiO2 of <200 mmHg with pulmonary edema on chest radiograph or use of ECMO.

SECONDARY OUTCOMES:
Number of patients with plasma EBV viral load of >=10,000 copies/mL | 12 months post-transplant
  Plasma EBV viral load of >=10,000 copies/mL. This will be compared to historic controls.

CONTACTS AND LOCATIONS:
Overall Officials: Deepali Kumar, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto General Hospital, Multi-Organ Transplant, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No